CLINICAL TRIAL: NCT02867449
Title: A Non-Inferiority Trial of Metacognitive Therapy Versus Exposure and Response Prevention for Individuals With Obsessive-Compulsive Disorder
Brief Title: Metacognitive Therapy for Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Philipps University Marburg (Other); German Research Foundation (Other)
Responsible Party: Principal Investigator, Cornelia Exner, Prof. Dr. Cornelia Exner, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCT_OCD
Record Dates: First submitted 2016-06-30; First posted 2016-08-16 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metacognitive Therapy (Experimental): Metacognitive Therapy for OCD according to Wells (1997)
  Interventions: Behavioral: Metacognitive Therapy
- Exposure and Response Prevention (Experimental): Exposure and Response Prevention for OCD according to Kozak & Foa (1997)
  Interventions: Behavioral: Exposure and Response Prevention

INTERVENTIONS:
Behavioral: Metacognitive Therapy — Metacognitive Therapy for OCD according to Wells (1997)
  Arms: Metacognitive Therapy
Behavioral: Exposure and Response Prevention — Exposure and Response Prevention for OCD according to Kozak & Foa (1997)
  Arms: Exposure and Response Prevention

SUMMARY:
Cognitive behavior therapy is the most effective treatment of obsessive-compulsive disorder. However, the majority of treated patients remain symptomatic. The metacognitive therapy by Wells (1997) could achieve substantial gains in first pilot studies. The purpose of this study is to investigate this approach with a randomized controlled trial by comparing metacognitive therapy with exposure and response prevention for obsessive-compulsive disorder.

DETAILED DESCRIPTION:
The purpose of this study is to investigate metacognitive therapy by Wells (1997) with a randomized controlled trial by comparing metacognitive therapy with exposure and response prevention for obsessive-compulsive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis: obsessive-compulsive disorder
* German-speaking
* Agreeing to participate, verified by completion of informed consent
* Stable medication (at least 4 weeks)

Exclusion Criteria:

* Current or past diagnosis of substance dependence, psychosis, neurological conditions
* Mental retardation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change in Symptom Severity (Yale Brown Obsessive-Compulsive Scale; Y-BOCS) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in Symptom Severity (Yale Brown Obsessive-Compulsive Scale; Y-BOCS)

SECONDARY OUTCOMES:
Change in Symptom Severity (Padua Inventory; PI) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in Symptom Severity (Padua Inventory; PI)
Change in general psychopathology (Symptom Checklist-90-Revised, SCL-90-R) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in general psychopathology (Symptom Checklist-90-Revised, SCL-90-R)
Change in Metacognitions (Metacognitions Questionnaire, short version, MCQ-30) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in Metacognitions (Metacognitions Questionnaire, short version, MCQ-30)
Change in Obsessive Beliefs (Obsessive Beliefs Questionnaire, OBQ) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in Obsessive Beliefs (Obsessive Beliefs Questionnaire, OBQ)
Change in Behavioral Avoidance (Behavioral Avoidance Test, BAT) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in Behavioral Avoidance (Behavioral Avoidance Test, BAT)
Change in Depression (Beck Depression Inventory, BDI-II) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in Depression (Beck Depression Inventory, BDI-II)
Change in Anxiety (Beck Anxiety Inventory, BAI) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in Anxiety (Beck Anxiety Inventory, BAI)
Change in Symptom Severity (Clinical Global Impressions; CGI) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in Symptom Severity (Clinical Global Impressions; CGI)
Change in psychosocial functioning (Global Assessment of Functioning Scale, GAF) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in psychosocial functioning (Global Assessment of Functioning Scale, GAF)
Change in quality of life (The World Health Organization Quality of Life, WHOQOL_BREF) | at pretest (admission), after completion of 6 therapeutic sessions (after an expected average of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected average of 12 weeks), at follow-up (6 months after end of treatment)
  Change in quality of life (The World Health Organization Quality of Life, WHOQOL_BREF)
Difference in efficiency (length of treatment) | immediately after completion of therapy (after an expected avarage of 12 weeks)
  documentation of number of sessions
Difference in medical costs (based on the length of treatment) | immediately after completion of therapy (after an expected avarage of 12 weeks)
  Difference in medical costs (based on the length of treatment)
Difference in negative effects of psychotherapy (Inventory for the Assessment of Negative Effects of Psychotherapy, INEP) | after completion of 6 therapeutic sessions (after an expected avarage of 6 weeks), at posttest after completion of 12 therapeutic sessions (after an expected avarage of 12 weeks), at follow-up (6 months after end of treatment)
  Difference in negative effects of psychotherapy (Inventory for the Assessment of Negative Effects of Psychotherapy, INEP)
Difference in satisfaction with the treatment | immediately after completion of therapy (after an expected avarage of 12 weeks)
  Difference in satisfaction with the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Exner, Prof. Dr., Principal Investigator — Leipzig University; Julia A. Glombiewski, Dr., Principal Investigator — Philipps University Marburg; Alexandra Kleiman, Dr., Study Director — Leipzig University; Anke Haberkamp, Dr., Study Director — Philipps University Marburg
Locations (2):
- Germany (2):
  - Leipzig University, Leipzig
  - Philipps University Marburg, Marburg

IPD SHARING:
Plan to Share IPD: Undecided